CLINICAL TRIAL: NCT06042920
Title: A Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Deucravacitinib in Participants With Non-Pustular PalmoPlantar and Genital Psoriasis (Psoriatyk Special Sites)
Brief Title: A Study to Evaluate Effectiveness and Safety of Deucravacitinib in Participants With Non-Pustular Palmoplantar and Genital Psoriasis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-1112; 2023-504663-16 (EudraCT Number); U1111-1289-6934 (Registry Identifier: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Palmoplantar Psoriasis; Genital Psoriasis
Keywords: Deucravacitinib; BMS-986165; SOTYKTU; Plaque psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo followed by Deucravacitinib (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165; SOTYKTU
Drug: Placebo — Specified dose on specified days
  Arms: Placebo followed by Deucravacitinib

SUMMARY:
The purpose of this study is to measure the safety and effectiveness of deucravatinib in participants with non-pustular palmoplantar psoriasis and genital psoriasis.

ELIGIBILITY:
Key Inclusion Criteria:

Inclusion Criteria for Non-Pustular Palmoplantar Psoriasis

* Men and women diagnosed with stable plaque psoriasis with involvement of the palm(s)and/or sole(s) for at least 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the investigator.
* Moderate-to-severe plaque psoriasis defined as s-PGA score of ≥ 3 on a 5-point scale at both screening visit and Day 1.
* Moderate-to-severe non-pustular PP psoriasis, defined as pp-PGA score of ≥ 3 on a 5-pointscale and pp-PASI ≥ 8 at both screening visit and Day 1.

  * A total maximum of 5 sterile pustules across both palms and soles limited only to psoriatic plaques will be allowed.
* Evidence of typical plaque psoriasis outside palms and soles at both screening visit and Day 1.
* Deemed by the investigator to be a candidate for phototherapy or systemic therapy.
* Failed to respond to, or intolerant of ≥ 1 topical therapy.

Inclusion Criteria for Genital Psoriasis

* Men and women diagnosed with stable plaque psoriasis with involvement of the genital area for at least 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the investigator.
* Moderate-to-severe plaque psoriasis defined as s-PGA score of ≥ 3 on a 5-point scale at both screening visit and Day 1.
* Moderate-to-severe GenPs, defined as static Physician's Global Assessment of Genitalia (s-PGA-G) score of ≥ 3 on a 6-point scale at both screening visit and Day 1.
* Evidence of typical plaque psoriasis in a non-genital area at both screening visit and Day 1.
* Deemed by the investigator to be a candidate for phototherapy or systemic therapy.
* Failed to respond to, or intolerant of ≥ 1 topical therapy.

Key Exclusion Criteria:

Target Disease Exceptions

* Has non-plaque psoriasis (for PP pustulosis, PP pustular psoriasis, isolated pustules on palms or soles with or without erythema outside psoriatic plaques, guttate, pustular, erythrodermic, and drug-induced psoriasis) at screening or Day 1.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With a 75% Improvement in Palmoplantar Psoriasis Area and Severity Index (pp-PASI-75) Score | Baseline to Week 16
Number of Participants With Static Physician Global Assessment Genitals (s-PGA-G) Score of 0 (Clear ) or 1 (Almost Clear), With At Least a 2-Point Reduction | Baseline to Week 16

SECONDARY OUTCOMES:
Number of Participants With Palmoplantar Physician Global Assessment (pp-PGA) Score of 0 (Clear) or 1 (Almost Clear), With At Least a 2-Point Reduction | Baseline to Week 16
Number of Participants With Static Physician Global Assessment (s-PGA) Score of 0 (Clear) or 1 (Almost Clear), With Least a 2-Point Reduction | Baseline to Week 16
Change from baseline in Genital Psoriasis (GenPs) Itch Numeric Rating Scale (NRS) score | Baseline to Week 16
Number of Participants With Adverse Events (AEs) | Up to Week 16
Number of Participants With Serious Adverse Events (SAEs) | Up to Week 16
Number of Participants With Clinical Laboratory Abnormalities | Up to Week 16
Number of Participants With Vital Sign Abnormalities | Up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (20):
  - Local Institution - 0050, Phoenix, Arizona
  - Local Institution - 0015, Fountain Valley, California
  - Local Institution - 0009, Los Angeles, California
  - Local Institution - 0004, Santa Monica, California
  - Local Institution - 0057, Skokie, Illinois
  - Local Institution - 0052, Indianapolis, Indiana
  - Local Institution - 0053, Plainfield, Indiana
  - Local Institution - 0029, Rockville, Maryland
  - Local Institution - 0012, Detroit, Michigan
  - Local Institution - 0005, East Windsor, New Jersey
  - Local Institution - 0002, New York, New York
  - Local Institution - 0008, New York, New York
  - Local Institution - 0062, New York, New York
  - Local Institution - 0001, Winston-Salem, North Carolina
  - Local Institution - 0066, Boardman, Ohio
  - Local Institution - 0055, Mayfield Heights, Ohio
  - Local Institution - 0056, Pittsburgh, Pennsylvania
  - Local Institution - 0010, Houston, Texas
  - Local Institution - 0007, Norfolk, Virginia
  - Local Institution - 0033, Mill Creek, Washington
- Argentina (4):
  - Local Institution - 0043, Ciudad Autónoma Buenos Aires, B
  - Local Institution - 0037, Ciudad Autónoma Buenos Aires, B
  - Local Institution - 0034, Ciudad Autonoma Buenos Aires, C
  - Local Institution - 0042, Rosario, S
- Canada (7):
  - Local Institution - 0058, Newmarket, Ontario
  - Local Institution - 0060, Toronto, Ontario
  - Local Institution - 0065, Montreal, Quebec
  - Local Institution - 0054, Montreal, Quebec
  - Local Institution - 0059, Québec, Quebec
  - Local Institution - 0061, Saint-Jérôme, Quebec
  - Local Institution - 0064, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol-Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.htm
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com